CLINICAL TRIAL: NCT01264393
Title: Using a State-Wide Initiative to Disseminate Effective Behavioral Weight Loss Strategies
Brief Title: State-wide Health Approach to Increase Reach and Effectiveness: Study 1
Acronym: SHARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rena R. Wing, Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2054-10; R18DK083248 (NIH)
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Shape Up Rhode Island + Online weight loss program + groups (Active Comparator): Participants assigned to this arm will receive the standard Shape Up Rhode Island statewide intervention, an internet-based weight loss program, and the option of attending face-to-face group sessions
  Interventions: Behavioral: Shape Up Rhode Island + Online Weight Loss Program + Group sessions
- Shape Up Rhode Island + Online Weight Loss Program (Active Comparator): Participants assigned to this arm will receive the standard Shape Up Rhode Island statewide intervention in addition to an internet-based weight loss program
  Interventions: Behavioral: Shape Up Rhode Island + Online Weight Loss Program
- Shape Up Rhode Island + Internet Resources (Active Comparator): Participants in this arm will receive the Standard Shape Up Rhode Island statewide intervention plus access to internet resources
  Interventions: Behavioral: Shape Up Rhode Island + Online Resources

INTERVENTIONS:
Behavioral: Shape Up Rhode Island + Online Resources — Participants will receive Shape Up Rhode Island, which is a 12-week statewide physical activity and weight loss campaign in addition to online weight loss resources
  Arms: Shape Up Rhode Island + Internet Resources
Behavioral: Shape Up Rhode Island + Online Weight Loss Program — Participants will receive Shape Up Rhode Island, a 12-week statewide physical activity and weight loss campaign in addition to an online weight loss program
  Arms: Shape Up Rhode Island + Online Weight Loss Program
Behavioral: Shape Up Rhode Island + Online Weight Loss Program + Group sessions — Participants will receive Shape Up Rhode Island, a 12-week statewide physical activity and weight loss campaign in addition to an online weight loss program and the option of attending group sessions
  Arms: Shape Up Rhode Island + Online weight loss program + groups

SUMMARY:
Behavioral weight loss programs can successfully reduce body weight, but these programs are available to limited numbers of overweight and obese individuals. This project evaluates a unique weight loss approach that combines a self-sustaining weight loss campaign (for outreach) with training in behavioral weight loss strategies and strategies to increase accountability (to improve weight loss success). This innovative combination has the potential to be a cost-effective model for disseminating weight control interventions.

DETAILED DESCRIPTION:
Participants will be randomly assigned to 1 of 3 treatment arms: Shape Up Rhode Island (SURI; a community-based weight loss campaign), SURI plus an Internet-based behavioral weight loss program (SURI + IBWL), or SURI + IBWL + optional group sessions (SURI + IBWL + Group). Primary outcome is weight loss at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 years
2. Body Mass Index >25 kg/m2
3. Both genders will be recruited; it is estimated that 70% of participants will be women.
4. All ethnic groups will be recruited, with a goal of recruiting 33% minorities (see below for specific recruitment plans)
5. No health problems that make weight loss or unsupervised exercise unsafe
6. English speaking

Exclusion criteria:

1. report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q; items 1-4). Individuals endorsing joint problems, prescription medication use or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
2. are currently pregnant or intend to become pregnant in the next 12 months
3. are planning to move outside of the state within the next 12 months
4. have previously participated in the Shape Up Rhode Island 2008 pilot study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Weight change from the initial assessment to the 3-month follow-up assessment measured on a digital scale to the nearest 0.1-kilogram. | 0 to 3 months

SECONDARY OUTCOMES:
Weight change from the initial assessment to the 6-month follow-up assessment measured on a digital scale to the nearest 0.1-kilogram. | 0 to 6 months
Weight change from the initial assessment to the 12-month follow-up assessment measured on a digital scale to the nearest 0.1-kilogram. | 0 to 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Rena R. Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Background] Wing RR, Crane MM, Thomas JG, Kumar R, Weinberg B. Improving weight loss outcomes of community interventions by incorporating behavioral strategies. Am J Public Health. 2010 Dec;100(12):2513-9. doi: 10.2105/AJPH.2009.183616. Epub 2010 Oct 21. PMID 20966375
- [Derived] Naparstek J, Wing RR, Xu X, Leahey TM. Internet-delivered obesity treatment improves symptoms of and risk for depression. Obesity (Silver Spring). 2017 Apr;25(4):671-675. doi: 10.1002/oby.21773. Epub 2017 Feb 22. PMID 28224713